CLINICAL TRIAL: NCT05299619
Title: A Prospective Study Assessing the Impact of Tixel Treatment of Peri-orbital Wrinkles on Dry Eye Symptoms and Signs in Patients With Dry Eye
Brief Title: Tixel Treatment for Dry Eye Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Ludger Hanneken (Other)
Responsible Party: Sponsor-Investigator, Dr Ludger Hanneken, Principle investigator, Vallmedic Vision & Aesthetic
Organization: Vallmedic Vision & Aesthetic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN0683
Record Dates: First submitted 2021-12-21; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Peri-orbital Wrinkles; Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: A single-center, prospective, non-masked, pilot study, to assess the safety and efficacy of the Tixel treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tixel Group (Experimental): Tixel treatments in Dry Eye Patients
  Interventions: Device: Tixel

INTERVENTIONS:
Device: Tixel — a thermomechanical system developed for fractional treatment. The system is designed for the treatment of soft tissue by direct conduction of heat, enabling fast water evaporation with low thermal damage to the surrounding tissue (such as charring or ablation).
  Other Names: thermomechanical system

SUMMARY:
Dry eye syndrome is caused by a chronic lack of sufficient lubrication and moisture on the surface of the eye. Consequences of dry eyes range from subtle but constant eye irritation to significant inflammation and even scarring of the front surface of the eye. Meibomian Gland Dysfunction (MGD) refers to the condition where the glands are not secreting enough oil or when the oil they secrete is of poor quality.

Tixel is a fractional skin rejuvenation system, which relies on direct thermal energy delivery, free of any radiation type such as laser, RF, etc. The energy is transferred via a continuously sterile, thermal titanium element (the "Tip"), located on the applicator (the "Handpiece"). In this study, the principal investigator will undertake standard treatment of periorbital wrinkles with Tixel and observe the effect on dry eye disease symptoms and signs.

DETAILED DESCRIPTION:
Tixel® (Novoxel®, Israel) is a thermomechanical system developed for fractional treatment. The system is designed for the treatment of soft tissue by direct conduction of heat, enabling fast water evaporation with low thermal damage to the surrounding tissue (such as charring or ablation). The system consists of a handpiece connected to a console. The handpiece applies a therapeutic element, the "tip", fixated on the distal section. The tip is comprised of a gold-plated copper base and a thin-walled titanium alloy cover.

While treating patients for wrinkles, it has been observed that in several cases, treatment had an effect on subjects who have been suffering from a pre-condition of dry eye disease. The effect was expressed mainly by increased tearing.

In this study, the principal investigator will undertake standard treatment of periorbital wrinkles with Tixel and observe the effect on dry eye disease symptoms and signs.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years
2. Mild to Moderate Periorbital wrinkles
3. OSDI score of at least 23
4. Noninvasive Tear film break up time (NIKBUT) ≤ 10 seconds
5. Willing and able to provide written informed consent.
6. Willing to participate in all study activities and instructions.

Exclusion Criteria:

1. Pregnancy and breastfeeding
2. Lesions in the periorbital area
3. Acute severe blepharitis
4. Acute conjunctivitis
5. Other concomitant anterior eye disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Safety, Device related AE frequency in the study | 8 months
  Any safety related event during the study will be recorded and analysed
NIBUT in Seconds | 8 months
  Non-Invasive Break Up Time

SECONDARY OUTCOMES:
Efficacy assessment - OSDI-Ocular Surface Disease Index Questionnaire changes from baseline | 8 months
  OSDI Score; 12 Questions; answers between 0-4; Total score calculated 0-100. Higher score means worst Dry Eye Symptomes
Osmolarity mOsml/L | 8 months
  Osmolarity test with TearLab
Staining; Total Ocular Staining Score | 8 month
  Corneal staining fluorescein and conjunctival/lid margin staining lissamine green

CONTACTS AND LOCATIONS:
Locations (1):
- Vallmedic Vision & Aesthetic, Les Escaldes, Andorra

IPD SHARING:
Plan to Share IPD: No